CLINICAL TRIAL: NCT06908525
Title: A Translation Study of the Things You Do Questionnaire 15-Item Version
Brief Title: Norwegian Translation of the Things You Do Questionnaire 15-Item Version
Acronym: TYDQ-15
Status: Not yet recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Aleksander Gulla Heltne, Principal Investigator, Haukeland University Hospital
Other Study IDs: 897112; 309264 (Other Grant/Funding Number: Research Council of Norway)
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: General Adult Population; Age 16 and Older
Keywords: Translation; TYDQ-15; Psychometric Evaluation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Psychotherapy aims to modify dysfunctional patterns of thinking, feeling, and behaving to improve mental health. A five-factor model of adaptive behaviors, operationalized in the Things You Do Questionnaire (TYDQ), has been identified as a mediator of treatment response in depression and anxiety interventions. The short-form TYDQ-15 is a key component of a transdiagnostic treatment promoting adaptive behavior. To implement this intervention in Norway, the TYDQ-15 requires translation and cultural adaptation, following established guidelines for clinical assessment instruments. Currently unavailable in Norwegian, its translation and psychometric evaluation are necessary for clinical application. This study aims to (1) produce a culturally adapted Norwegian version of the TYDQ-15 and (2) assess its psychometric properties, including reliability, factor structure, and criterion validity, within a Norwegian population. The findings will facilitate the integration of the Things You Do Intervention into Norwegian mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Native Norwegian speaker

Exclusion Criteria:

* Does not speak Norwegian fluently

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population of Norway
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Things You Do Questionnaire 15-Item Version (TYDQ-15) | Singe time point, at enrolment.
  The Things You Do Questionnaire - 15 Item Version (TYDQ-15) measures how frequently one engages in adaptive behavior with 15 items scored 0 ("never") to 4 ("every day"). The 15 items are grouped into the five domains of "meaningful activities", "healthy thinking", "goals and plans", "healthy routines", and "social connections. The original English language instrument has been shown to have acceptable psychometric properties across representative population samples.

SECONDARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9) | Single time point, at enrolment.
  The Patient Health Questionnaire (PHQ-9) - measures depression severity with nine items scored 0 ("not at all") to 3 ("nearly every day"), corresponding to the criteria for major depression in the DSM-5. The sum of the nine items ranges from 0-27. The scale has demonstrated adequate psychometric properties across different samples and has been found to be sensitive to change in depressive symptoms.
The Generalized Anxiety Disorder Scale (GAD-7) | Single time point, at enrolment.
  The Generalized Anxiety Disorder Scale (GAD-7) - measures anxiety severity with seven items scored 0 ("not at all") to 3 ("nearly every day") corresponding to symptoms of anxiety disorders. The sum score ranges from 0-21. GAD-7 has demonstrated adequate psychometric properties across different samples and has been found to be sensitive to the presence of anxiety disorders.
The Satisfaction with Life Scale (SWLS) | Single time point, at enrolment.
  The Satisfaction with Life Scale (SWLS) - measures life-satisfaction with 5 items scored 1 ("strongly disagree") to 7 ("strongly agree"), corresponding to statements of general life satisfaction. Sum scores range from X to Y with higher scores indicating greater life satisfaction. The SWLS has demonstrated adequate psychometric properties across different samples.

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of IPD for this study will require guaranteed anonymity for all involved participants. Unless such anonymity can be guaranteed, IPD will not be shared outside the research team. Current advances in machine learning and AI introduce difficult questions regarding the possibility of re-identification of research participants from patterns in the data. Decisions of IPD publication therefore require additional consideration.